CLINICAL TRIAL: NCT04114864
Title: A Primary Prevention Intervention for the Promotion of Psycho-social Wellbeing in Adolescent Young Carers: a Randomized Control Trial in the Project H2020 ME-WE
Brief Title: A Primary Prevention Intervention for the Promotion of Psycho-social Wellbeing in Adolescent Young Carers:
Acronym: ME-WE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Valentina Hlebec (Other)
Collaborators: LINNEUNIVERSITETET (LNU), Sweden (leading the consortium) (Unknown); EUROCARERS-ASSOCIATION EUROPEENNE TRAVAILLANT AVEC ET POUR LES (Unknown); THE UNIVERSITY OF SUSSEX (UoS), UK (Unknown); CARERS TRUST (Carers Trust), UK (Unknown); STIFTUNG KALAIDOS FACHHOCHSCHULE (Kalaidos FH), SW (Unknown); MINISTERIE VAN VOLKSGEZONDHEID, WELZIJN EN SPORT (NLNA), NL (Unknown); STICHTING VILANS (VILANS), NL (Unknown); ISTITUTO NAZIONALE DI RIPOSO E CURA PER ANZIANI INRCA (INRCA), IT (Unknown); ANZIANI E NON SOLO SOCIETA COOPERATIVA SOCIALE (ANZIANI E), IT (Unknown); UNIVERZA V LJUBLJANI (UL), SI (Unknown); Nationellt kompetenscentrum anhöriga (Nka), (Swedish Family Care Competence Centre), Kalmar, Sweden (Unknown)
Responsible Party: Sponsor-Investigator, Valentina Hlebec, prof. dr. Valentina Hlebec; wp6 leader, University of Ljubljana
Organization: University of Ljubljana (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 754702
Record Dates: First submitted 2019-09-22; First posted 2019-10-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Adolescent - Emotional Problem; Mental Health Wellness 1; Caregivers; Primary Prevention; Cognitive Therapy
Keywords: Adolescent; Acceptance and Commitment Therapy, Cognitive therapy; Mindfulness; Europe

STUDY DESIGN:
Intervention Model Description: The study is a prospective C-RCT, with a two (group) by three (time) repeated measures factorial design. Both the intervention and the wait-list control group will be assessed at baseline, immediately post-intervention for the intervention group or after 7 weeks for the wait-list control group - and at the 3MFU.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): This arm will be receiving the 7 ME-WE sessions psycho-educational intervention. The experimental group will involve a blended approach with 'face to face' meetings in three European partner countries and online sessions (via a ME-WE mobile app) and a purely 'f2f' approach in a further three European partner countries.
  Interventions: Behavioral: Psycho-educational sessions
- Control (Placebo Comparator): The control-group will be a wait-list, receiving relaxation exercises during waiting.
  Interventions: Behavioral: Psycho-educational sessions

INTERVENTIONS:
Behavioral: Psycho-educational sessions — Participants of clusters allocated to the ME-WE intervention group will complete a programme based on seven weekly sessions of approximately 2 hours each, plus a follow-up meeting after 3 months from the end of the programme. All sessions maintain a similar structure (objectives, ice-breaker, central activity/ies, and final activity). At the end of some sessions, participants will be asked to do some exercises at home, between one meeting and the next one, in order to keep what has been done during the previous session fresh in their minds.
  Contents of sessions will be as follows: (1) Getting to know each other; (2) The Advisor: dealing with annoying thoughts; (3) The Noticer: being in connection with our feelings; (4) The Discoverer: growing and thriving; (5) Values: connecting to meaning and vitality; (6) Developing a flexible self-view and self-compassion; (7) Building strong social networks.
  Other Names: Acceptance and Commitment Therapy - Mental Health- Mindfulness

SUMMARY:
Adolescent young carers (AYCs) are young people aged 15-17 years old, who take on significant or substantial caring tasks and assume a level of responsibility that would usually be associated with an adult. In Europe, the estimated prevalence rate of YCs is around 4-8%.Taking on care responsibilities so early in life may have considerable negative consequences for YCs' mental and physical health and psychosocial development. Psychosocial interventions to support YC worldwide are generally quite limited. The H2020 Me-We project (Psychosocial Support for Promoting Mental Health and Well-being among Adolescent Young Carers in Europe) aims to develop an innovative framework of primary prevention interventions for adolescent YCs (AYCs) aged 15-17 to be tested in six European countries (Italy, Netherlands, Slovenia, Sweden, Switzerland, United Kingdom).

The theoretical framework chosen for the intervention is the DNA-V Model. The DNA-V model is a psychological intervention, addressed to adolescents and young people, used in educational and clinical settings. This model has its roots in the contextual and functional science and it is based on Acceptance and Commitment Therapy, a third-generation cognitive-behavioural therapy. The intervention programme designed for the ME-WE project builds on the DNA-V model but it was adapted to fit the specific needs of adolescent young carers (AYCs) and the goals of the ME-WE project.

The study aim is to evaluate the efficacy of DNA-V based program for AYCs (so-called ME-WE intervention), using a cluster-randomized controlled trial (C-RCT) design. The evaluation of the intervention will be carried out using as primary outcome variables: Psychological flexibility; Mindfulness skills; Resilience; Subjective mental health; Quality of life; Subjective health complaints; Caring-related quality of life; Cognitive and emotional impact of caring and Social support. As secondary outcome variables will be included Self-reported school, training or work experience, performance, and attendance.

COVID-19 Amendment: Recruitment, should be moved to a cluster- based online recruitment or individual, social media recruitment, face-to-face sessions should be moved to online sessions using video-conferencing instruments, allowing for visual presentations of participants and session materials (e.g. ZOOM, Microsoft Teams). Four open-ended items were added to evaluation questionnaire assessing impact of COVID-19 pandemic.

DETAILED DESCRIPTION:
Adolescent young carers (AYCs) are young people aged 15-17 years old, who take on significant or substantial caring tasks and assume a level of responsibility that would usually be associated with an adult. Often on a regular basis, they look after family member(s) with a disability, chronic physical and/or mental health condition or substance use issue and/or problems related to old age, who require support or supervision. In Europe, the estimated prevalence rate of YCs is around 4-8%.

Taking on care responsibilities so early in life may have considerable negative consequences for YCs' mental and physical health and psychosocial development. Furthermore, YCs likely face difficulties in education that negatively impact their future employability and socio-economic status and experience constraints in finding and maintaining employment and pursuing their career aspirations.

Psychosocial interventions to support YC worldwide are generally quite limited. In order to prevent the entrenched level of caring that results in significant and long-term effects on YCs' well-being and hinder transitions to adulthood, it has been suggested that a primary prevention model should be adopted. To prevent adverse mental health, social, and educational outcomes in YCs, building their resilience would be especially important.

The H2020 Me-We project (Psychosocial Support for Promoting Mental Health and Well-being among Adolescent Young Carers in Europe) aims to develop an innovative framework of primary prevention interventions for adolescent YCs (AYCs) aged 15-17 to be tested in six European countries (Italy, Netherlands, Slovenia, Sweden, Switzerland, United Kingdom).

The theoretical framework chosen for the intervention is the DNA-V Model. The DNA-V model is a psychological intervention, addressed to adolescents and young people, used in educational and clinical settings. This model has its roots in the contextual and functional science and it is based on Acceptance and Commitment Therapy, a third-generation cognitive-behavioural therapy. The intervention programme designed for the ME-WE project builds on the DNA-V model but it was adapted to fit the specific needs of adolescent young carers (AYCs) and the goals of the ME-WE project.

The study aim is to evaluate the efficacy of DNA-V-based program for AYCs, called the ME-WE support intervention, using a cluster-randomized controlled trial (C-RCT) design. The evaluation of the intervention will be carried out using as primary outcome variables: Psychological flexibility; Mindfulness skills; Resilience; Subjective mental health; Quality of life; Subjective health complaints; Caring-related quality of life; Cognitive and emotional impact of caring and Social support. As secondary outcome variables Self-reported school, training or work experience, performance, and attendance will be used. Control variable will be caring activities; overall amount of caring and likes and dislikes about caring. Results will be compared of the intervention-group participants relative to the wait-list control-group participants from baseline (pre-intervention) through post-intervention and 3-month follow-up (3MFU).

Investigators expect that there will be greater improvements in protective factors targeted by the ME-WE intervention. Thus, it is hypothesized that, compared to the wait-list control group, ME-WE participants will report greater improvements in psychological flexibility, mindfulness, resilience, subjective mental health and quality of life as well as in perceived emotional impact of caring and social support (primary outcomes), and these effects will be maintained at the 3MFU. The impact of ME-WE on self-reported school, training or work experience, performance, and attendance of AYCs (secondary outcomes) will be also explored. Since the intervention will not address these variables directly, we consider them as secondary outcomes.

COVID-19 Amendment: Recruitment, should be moved to a cluster- based online recruitment or individual, social media recruitment, face-to-face sessions should be moved to online sessions using video-conferencing instruments, allowing for visual presentations of participants and session materials (e.g. ZOOM, Microsoft Teams). All evaluation self-report instruments are available online. Five open-ended items were added to evaluation questionnaire assessing impact of COVID-19 pandemic (how participants were affected by pandemic, what kind of support and services they received, how their mental and/or physical health has been affected and how they experience the participation in intervention).

ELIGIBILITY:
Inclusion Criteria:

1. being between 15 and 17 years of age;
2. taking on caring tasks for family member(s) (e.g., parents, siblings, grandparents) with a disability, chronic physical and/or mental health condition or substance use issue and/or problems related to old age (Becker, 2000; Metzing-Blau & Schnepp, 2008).

Exclusion Criteria:

1. Concurrently participating in other psychotherapies or mindfulness-based interventions/ programmes;
2. Having started a new psychotropic medication within the past 30 days or planning on starting or changing psychotropic medication during the course of the study;
3. limited knowledge of local language (in all countries except Sweden)..

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 295 (Actual)
Dates: Start 2019-10-20 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Psychological flexibility at 5 months | baseline, end (after about 7 weeks), follow up after 3 months from completion
  Avoidance and fusion questionnaire for youth (AFQ-Y; Greco, Lambert, & Baer, 2011); 8 items on a 5-point scale (from 'not at all true' to 'very true'), overall total score.
Change from baseline Mindfulness skills at 5 months | baseline, end (after about 7 weeks), follow up after 3 months from completion
  Child and Adolescent Mindfulness Measure (CAMM; Greco, Baer, & Smith, 2011); 10 items on a 5-point scale (from 'never true' to 'always true'), overall total score.
Change from baseline Resilience at 5 months | baseline, end (after about 7 weeks), follow up after 3 months from completion
  Brief Resilience Scale (BRS; Smith 2008); six items on a 5-point Likert scale (from 'strongly disagree' to 'strongly agree'), overall total score.
Change from baseline Subjective mental health at 5 months | baseline, end (after about 7 weeks), follow up after 3 months from completion
  Warwick Edinburgh Mental Well-Being Scale (WEMWBS; Tennant et al., 2007); 14 items on a 5-point Likert scale ('none of the time', 'rarely', 'some of the time', 'often', 'all of the time'), overall total score.
Change from baseline Quality of life at 5 months | baseline, end (after about 7 weeks), follow up after 3 months from completion
  Kidscreen 10 (RavensSieberer, & the KIDSCREEN Group Europe, 2006); 10 items on 5-point Likert scale from 'not at all / never' to 'extremely / always'; one global health-related quality of life score.
Change from baseline Subjective health complaints at 5 months | baseline, end (after about 7 weeks), follow up after 3 months from completion
  HBSC Symptom Checklist (HBSC-SCL); 8 items on a 5-point scale ('rarely or never', 'almost every month', 'more than once par week', 'almost every week', 'almost every day').
Change from baseline Caring-related quality of life at 5 months | baseline, end (after about 7 weeks), follow up after 3 months from completion
  Closed ended, ad hoc questions regarding thoughts about hurting themselves/others; being bullied, teased or made fun of; and experiencing some health-related issues because of their caring role.
Change from baseline Cognitive and emotional impact of caring at 5 months | baseline, end (after about 7 weeks), follow up after 3 months from completion
  Positive and Negative Outcomes of Caring (PANOC; Joseph et al., 2009; Joseph, Becker, & Becker, 2012); 20 items on a 3-point scale: 'never', 'some of the time' and 'a lot of the time'; two scores: positive and negative outcomes.
Change from baseline Social support at 5 months | baseline, end (after about 7 weeks), follow up after 3 months from completion
  : Brief Social Support Questionnaire (BSSQ; Sarason, Sarason, Shearin, & Pierce et al., 1987); 6 items with number of support sources as the response option.

SECONDARY OUTCOMES:
Change from baseline Self-reported school, training or work experience, performance, and attendance at 5 months | baseline, end (after about 7 weeks), follow up after 3 months from completion
  Closed ended, ad hoc questions regarding current education, training, or work, experiencing difficulties and effect of caring.
  Two open ended questions with a number of days as a response option (days being late or missed at school, training or work because of caring in the last 2 weeks of term time).

OTHER OUTCOMES:
Control variables: 1) Caring activities | baseline, end (after about 7 weeks), follow up after 3 months from completion
  1) Caring activities: Multidimensional Assessment of Caring Activities (MACA-YC18; Joseph, Becker, Becker, & Regel, 2009); 18 items on a 3-point scale: 'never', 'some of the time' and 'a lot of the time'; total score and six subscale scores for domestic tasks, household management, personal care, emotional care, sibling care, and financial/ practical care.
2) Overall amount of caring | baseline, end (after about 7 weeks), follow up after 3 months from completion
  Two open ended ad hoc questions with a number of hours as a response option (hours or caring per week for a typical day during week and at the weekend)
3) Likes and dislikes about caring | baseline, end (after about 7 weeks), follow up after 3 months from completion
  Three open ended, ad hoc questions regarding which one of their caring jobs they like the most, dislike the most or it upsets them the most?
Process evaluation outcomes (for intervention group only): | follow up after 3 months from completion
  - Post Intervention Self-Assessment adapted for the present study (PISA-CT2012; Joseph et al., 2009). Five open ended questions regarding e.g. the help and support they have been getting from the intervention, things that have changed for them because of attending this project, things they liked or didn't like about attending the project.
Process evaluation outcomes | end (if applicable), follow-up after 3 months from completion
  Four open ended items evaluating COVID-19 impact on participants

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Hanson, PhD Nursing, Principal Investigator — Linneus University, Kalmar, Sweden
Locations (6):
- Anziani e non solo soc. coop. soc, Carpi, Italy
- Stichting Vilans, Utrecht, Netherlands
- University of Ljubljana, Ljubljana, Slovenia
- Linnaeus University, Nationellt kompetenscentrum anhöriga (Nka), (Swedish Family Care Competence Centre), Kalmar, Sweden
- Stiftung Kalaidos Fachhochschule (Kalaidos FH), Zurich, Switzerland
- Carers Trust, Print Rooms, 164-180 Union Street, London, SE1 0LN. Carers Trust will be co-ordinating the completion of the interventions for the clinical trials in the UK. All trials for the ME-WE project will be completed in England., London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized evaluation data to be stored in data archive with limited access.
Supporting Information: Study Protocol
Time Frame: After the completion of the project, but the date is unknown.
Access Criteria: not yet known

REFERENCES:
- [Background] Acton, J., & Carter, B. (2016). The impact of immersive outdoor activities in local woodlands on young carers emotional literacy and well-being. Comprehensive Child and Adolescent Nursing, 39(2), 94-106.
- [Background] Aldridge, J. (2018). Where are we now? Twenty-five years of research, policy and practice on young carers. Critical Social Policy, 38(1), 155-165.
- [Background] Assaf RR, Auf der Springe J, Siskowski C, Ludwig DA, Mathew MS, Belkowitz J. Participation Rates and Perceptions of Caregiving Youth Providing Home Health Care. J Community Health. 2016 Apr;41(2):326-33. doi: 10.1007/s10900-015-0100-7. PMID 26483035
- [Background] Becker, S. (2000). Young carers. In M. Davies (Ed.), The Blackwell encyclopedia of social work (3rd ed.). Oxford: Blackwell.
- [Background] Becker, S. (2007). Global perspectives on children's unpaid caregiving in the family: Research and policy on 'young carers' in the UK, Australia, the USA and Sub-Saharan Africa. Global Social Policy, 7(1), 23-50.
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546
- [Background] Cohen, J. (1988). Statistical Power Analysis for the Behavioral Sciences (2nd ed.). Hillsdale, NJ: Erlbaum.
- [Background] Cunningham, L. C., Shochet, I. M., Smith, C. L., & Wurfl, A. (2017). A qualitative evaluation of an innovative resilience-building camp for young carers. Child & Family Social Work, 22(2), 700-710.
- [Background] Daniel, W. W. (1999). Biostatistics: A foundation for analysis in the health sciences (7th ed.). New York: John Wiley and Sons.
- [Background] Fraser E, Pakenham KI. Evaluation of a resilience-based intervention for children of parents with mental illness. Aust N Z J Psychiatry. 2008 Dec;42(12):1041-50. doi: 10.1080/00048670802512065. PMID 19016092
- [Background] Gettings S, Franco F, Santosh PJ. Facilitating support groups for siblings of children with neurodevelopmental disorders using audio-conferencing: a longitudinal feasibility study. Child Adolesc Psychiatry Ment Health. 2015 Apr 7;9:8. doi: 10.1186/s13034-015-0041-z. eCollection 2015. PMID 25866558
- [Background] Greco LA, Baer RA, Smith GT. Assessing mindfulness in children and adolescents: development and validation of the Child and Adolescent Mindfulness Measure (CAMM). Psychol Assess. 2011 Sep;23(3):606-14. doi: 10.1037/a0022819. PMID 21480722
- [Background] Greco LA, Lambert W, Baer RA. Psychological inflexibility in childhood and adolescence: development and evaluation of the Avoidance and Fusion Questionnaire for Youth. Psychol Assess. 2008 Jun;20(2):93-102. doi: 10.1037/1040-3590.20.2.93. PMID 18557686
- [Background] Schlarmann JG, Metzing S, Schoppmann S, Schnepp W. Germany's First Young Carers Project's Impact on the Children: Relieving the Entire Family. A Qualitative Evaluation. Open Nurs J. 2011;5:86-94. doi: 10.2174/1874434601105010086. Epub 2011 Oct 26. PMID 22135716
- [Background] Halliburton, A. E., & Cooper, L. D. (2015). Applications and adaptations of Acceptance and Commitment Therapy (ACT) for adolescents. Journal of Contextual Behavioral Science, 4(1), 1-11.
- [Background] Hamilton, M. G., & Adamson, E. (2013). Bounded agency in young carers' lifecourse-stage domains and transitions. Journal of Youth Studies, 16(1), 101-117.
- [Background] Hamilton, M., & Cass, B. (2017). Capturing the centrality of age and life-course stage in the provision of unpaid care. Journal of Sociology, 53(1), 79-93.
- [Background] Harris, R. (2009). ACT made simple: An easy-to-read primer on Acceptance and Commitment Therapy. Oakland, CA: New Harbinger.
- [Background] Hayes, L., & Ciarrochi, J. (2015). The Thriving Adolescent: Using acceptance and commitment therapy and positive psychology to help teens manage emotions, achieve goals, and build positive connections. Oakland, CA: New Harbinger.
- [Background] Hayes, S., Wilson, K., & Strosahl, K. (1999). Acceptance and commitment therapy: An experiential approach to behavior change. New York: Guilford.
- [Background] Heyman, A. (2013). Partnership working between young carers project and social services. Social Work and Social Sciences Review, 16(3), 50-64.
- [Background] Heyman, A., & Heyman, B. (2013). 'The sooner you can change their life course the better': The time-framing of risks in relationship to being a young carer. Health, Risk & Society, 15(6-7), 561-579.
- [Background] Järkestig-Berggren, U., Bergman, A. S., Eriksson, M., & Priebe, G. (2018). Young carers in Sweden-A pilot study of care activities, view of caring, and psychological well-being. Child & Family Social Work.
- [Background] Joseph S, Becker S, Becker F, Regel S. Assessment of caring and its effects in young people: development of the Multidimensional Assessment of Caring Activities Checklist (MACA-YC18) and the Positive and Negative Outcomes of Caring Questionnaire (PANOC-YC20) for young carers. Child Care Health Dev. 2009 Jul;35(4):510-20. doi: 10.1111/j.1365-2214.2009.00959.x. Epub 2009 Mar 23. PMID 19320904
- [Background] Joseph S, Kendall C, Toher D, Sempik J, Holland J, Becker S. Young carers in England: Findings from the 2018 BBC survey on the prevalence and nature of caring among young people. Child Care Health Dev. 2019 Jul;45(4):606-612. doi: 10.1111/cch.12674. Epub 2019 May 24. PMID 30995694
- [Background] Kallander, E. K., Weimand, B., Ruud, T., Becker, S., Van Roy, B., & Hanssen-Bauer, K. (2018). Outcomes for children who care for a parent with a severe illness or substance abuse. Child & Youth Services. https://doi.org/10.1080/0145935X.2018.1491302
- [Background] Kallapiran K, Koo S, Kirubakaran R, Hancock K. Review: Effectiveness of mindfulness in improving mental health symptoms of children and adolescents: a meta-analysis. Child Adolesc Ment Health. 2015 Nov;20(4):182-194. doi: 10.1111/camh.12113. Epub 2015 Sep 8. PMID 32680348
- [Background] Leu, A., Frech, M., Wepf, H., Sempik, J., Joseph, S., Helbling, L., ... & Jung, C. (2018). Counting young carers in Switzerland - A study of prevalence. Children & Society. https://doi.org/10.1111/chso.12296
- [Background] Leu, A., & Becker, S. (2017). A cross-national and comparative classification of in-country awareness and policy responses to 'young carers'. Journal of Youth Studies, 20(6), 750-762.
- [Background] Lloyd, K. (2013). Happiness and well-being of young carers: Extent, nature and correlates of caring among 10 and 11 year old school children. Journal of Happiness Studies, 14(1), 67-80.
- [Background] Merry SN, Hetrick SE, Cox GR, Brudevold-Iversen T, Bir JJ, McDowell H. Psychological and educational interventions for preventing depression in children and adolescents. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD003380. doi: 10.1002/14651858.CD003380.pub3. PMID 22161377
- [Background] Metzing-Blau S, Schnepp W. Young carers in Germany: to live on as normal as possible - a grounded theory study. BMC Nurs. 2008 Dec 24;7:15. doi: 10.1186/1472-6955-7-15. PMID 19108719
- [Background] Nagl-Cupal M, Daniel M, Koller MM, Mayer H. Prevalence and effects of caregiving on children. J Adv Nurs. 2014 Oct;70(10):2314-25. doi: 10.1111/jan.12388. Epub 2014 Mar 24. PMID 24660847
- [Background] Petts, R. A., Duenas, J. A., & Gaynor, S. T. (2017). Acceptance and Commitment Therapy for adolescent depression: Application with a diverse and predominantly socioeconomically disadvantaged sample. Journal of Contextual Behavioral Science, 6(2), 134-144.
- [Background] Purcal, C., Hamilton, M., Thomson, C., & Cass, B. (2012). From assistance to prevention: Categorizing young carer support services in Australia, and international implications. Social Policy & Administration, 46(7), 788-806.
- [Background] Sarason, I. G., Sarason, B. R., Shearin, E. N., & Pierce, G. R. (1987). A brief measure of social support: Practical and theoretical implications. Journal of Social and Personal Relationships, 4(4), 497-510.
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Stamatopoulos, V. (2016). Supporting young carers: a qualitative review of young carer services in Canada. International Journal of Adolescence and Youth, 21(2), 178-194.
- [Background] Swain, J., Hancock, K., Dixon, A., & Bowman, J. (2015). Acceptance and commitment therapy for children: A systematic review of intervention studies. Journal of Contextual Behavioural Science, 4, 73-85.
- [Background] Swain, J., Hancock, K., Hainsworth, C., & Bowman, J. (2015). Mechanisms of change: Exploratory outcomes from a randomised controlled trial of acceptance and commitment therapy for anxious adolescents. Journal of Contextual Behavioral Science, 1(4), 56-67.
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Derived] Hanson E, Barbabella F, Magnusson L, Brolin R, Svensson M, Yghemonos S, Hlebec V, Bolko I, Boccaletti L, Casu G, Hoefman R, de Boer AH, de Roos S, Santini S, Socci M, D'Amen B, Van Zoest F, de Jong N, Nap HH, de Jong Y, Bouwman T, Lewis F, Parkhouse T, Leu A, Phelps D, Guggiari E, Morgan V, Centola F, Joseph S, Becker S. Research and Innovation for and with Adolescent Young Carers to Influence Policy and Practice-The European Union Funded "ME-WE" Project. Int J Environ Res Public Health. 2022 Aug 11;19(16):9932. doi: 10.3390/ijerph19169932. PMID 36011572
- [Derived] Casu G, Hlebec V, Boccaletti L, Bolko I, Manattini A, Hanson E. Promoting Mental Health and Well-Being among Adolescent Young Carers in Europe: A Randomized Controlled Trial Protocol. Int J Environ Res Public Health. 2021 Feb 19;18(4):2045. doi: 10.3390/ijerph18042045. PMID 33669796